CLINICAL TRIAL: NCT03313882
Title: Na+ Channel mRNA Regulation in Heart Failure
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: Study00001184
Record Dates: First submitted 2017-08-31; First posted 2017-10-18 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure
Keywords: RNA Stability; HuR protein; SCN5A
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- donor: donor: normal heart samples from donor
  Interventions: Other: no intervention is involved
- ICM: ICM: heart samples with ischemic cardiomyopathy
  Interventions: Other: no intervention is involved
- NICM: NICM: heart samples with non-ischemic cardiomyopathy
  Interventions: Other: no intervention is involved

INTERVENTIONS:
Other: no intervention is involved

SUMMARY:
Human heart failure (HF) has been associated with reduced cardiac sodium channel current and other electrical remodeling. Recently, the investigators have shown that downregulation of cardiac Na+ channels (SCN5A) can contribute to arrhythmic risk and that upregulation can mitigate that risk. Furthermore, the investigators have shown that the reduction in cardiac SCN5A mRNA abundance is reflected in circulating white blood cells (WBCs), which also express SCN5A, and that a reduction in SCN5A is highly predictive of appropriate implanted cardiac defibrillator (ICD) therapy. These data suggest that SCN5A regulation contributes to arrhythmic risk in HF. Other electrical remodeling events thought to contribute to arrhythmic risk include reductions in K+ currents, including Ito, IK1 and IKs are responsible. These current reductions have been linked to reduced transcription, translation and expression of the corresponding channel subunits, such as Kv4.3, Kir2.1, KvLQT1, and accessory proteins including minK and K+ channel interacting protein 2. That all these ion channels are downregulated may suggest a common mechanism to reduce ion channel expression. In this application, the investigators intend to explore an entirely novel mechanism by which SCN5A and other ion channel mRNA abundances are reduced in HF.

DETAILED DESCRIPTION:
Altered gene expression has been traditionally focused on transcriptional regulation. Nevertheless, recent large-scale analyses have revealed that as many as half of all changes in the amounts of mRNA in responses to cellular signals can be attributed to altered rates of mRNA decay. In preliminary data, we show that HuR, a member of a class of RNA stabilizing proteins that bind to AU-rich elements (ARE), is expressed in the heart and contributes to Na+ channel mRNA stability by binding to SCN5A transcript. Furthermore, HuR appears to be downregulated in human HF, perhaps contributing to the downregulation of ion channels and increased arrhythmic risk seen in HF. We propose that HuR is downregulated in HF, that this downregulation contributes to reduced Na+ and other currents and increased arrhythmic risk, and that upregulation of HuR will reduce ion channel downregulations and arrhythmic risk in HF. The investigators specific aims are:

Aim 1: Determine the extent to which HuR can regulate ion currents in cardiomyocytes.

Aim 2: Determine the relative contributions of known ion channel posttranscriptional control mechanisms.

Aim 3: Determine the mechanism and extent to which HuR activity is downregulated in ischemic and nonischemic cardiomyopathy and the correlation with ion channel mRNA, protein, and current.

Aim 4: Determine the extent to which overexpression of HuR can raise ion channel mRNA, raise ion channel current, and reduce arrhythmic risk in ischemic and nonischemic cardiomyopathy.

Please be notified that only Aim 2 involves the usage of de-identified human heart samples.

ELIGIBILITY:
Inclusion Criteria:

* ischemic or non-ischemic cardiomyopathy Healthy Donor heart

Exclusion Criteria: N/A

* Not diagnosed with ischemic or non-ischemic cardiomyopathy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: heart samples from healthy donor or from patients with ischemic or non-ischemic cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
ion channel expression | Baseline
  mRNA and protein levels of cardiac ion channels, cardiac ion currents

SECONDARY OUTCOMES:
HuR change | Baseline
  mRNA, protein, phosphorylation, cleavage products, and localization

IPD SHARING:
Plan to Share IPD: No